CLINICAL TRIAL: NCT04559542
Title: Management of Body Weight Regulation, Symptoms of Low Energy Availability, Body Acceptance, Eating Disorders, and Sexual Harassment Among Female Martial Art Athletes, and Impact of COVID-19 on Training and Sport Participation
Brief Title: Body Weight Regulation, Disordered Eating Behaviour, and Experiences of Sexual Harassment in Female Martial Art Athletes
Acronym: FMAB
Status: Completed | Type: Observational
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Ostfold University College (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Professor Jorunn Sundgot-Borgen, Professor, Norwegian School of Sport Sciences
Other Study IDs: 20/00378
Record Dates: First submitted 2020-08-25; First posted 2020-09-23 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Body Weight Changes; Eating Disorder Symptom; Sexual Harassment; Covid19; RED S
Keywords: Mental health; Eating disorders; female athletes; physical health; Body dissatisfaction; Body acceptance; body weight
MeSH Terms: conditions — Body Weight Changes; Sexual Harassment; COVID-19; Relative Energy Deficiency in Sport; Psychological Well-Being; Feeding and Eating Disorders; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female material art athletes: Females practicing material art during recruitment time, in Oslo-area in Norway

SUMMARY:
Athletes in martial arts compete in categories separated by body weight, hence, many athletes need to adjust their habitual body weight during periods with competition preparation. Athletes competing in weight sensitive sports are previously identified with an increased risk for symptoms of low energy availability and of disordered eating. The methods used for body weight regulation are varied, and athletes without professional competent support, are prone to rely on harmful methods. And of importance, female athletes respond more negatively to attempts of body weight reduction with regards to health effects.

Athletes of martial art are not surrounded by the same professional competence seen in other organized sports within the international sport federations, and specifically health competence is lacking. Additionally, numbers of females competing in martial art have increased the last decade, but they still practice in a sport culture dominated by males; both with reference to the high number of male participants, and with reference to the coaches within this sport. Sports involving practice in intimate, physical interaction with coaches or opposing athletes, and in sports where clothing is minimal, may be a high risk of experiences of sexual harassment. There have been a few reports on harmful methods of body weight regulation within martial arts, however, little knowledge exists on the practice by female martial art athletes, and the related health effects. Information on experiences of sexual harassment have been sparse in sport generally, with very little knowledge from sports like martial arts specifically. This study aims to explore the practice of female martial art athletes on body weight regulation, recovery strategies, their body acceptance and symptoms of eating disorders, and any experiences of sexual harassment. Additionally, with regards to the recent onset of the Covid-19 pandemic, this study also explores the related experiences by the athletes on training- and eating routines.

DETAILED DESCRIPTION:
Low energy availability is a situation triggered by a low energy intake relatively to the total energy needs. It may typically occur when energy expenditure is increased by sporting activities concurrently to an unconscious or voluntarily insufficient increase in energy intake. This may cause a condition called Relative energy deficiency in sport (RED-s), indicating a high risk for several negative health effects and performance deterioration. Athletes competing in body weight sensitive sports or sports categorized by body weight, have been identified with higher prevalence of RED-s, and specifically young females. Although it is the total difference between energy needs and energy availability that causes such scenario, the methods used to regulate body weight do also matter. Athletes without proper guidance on nutritional needs, recovery strategies, and optimal body weight regulation have previously reported use of harmful dieting methods, like purging methods, dehydration methods, and use of pharmaceuticals. Thus, young females competing in weight sensitive sport, not receiving any professional health and performance coaching are at specific risk for acutely and longterm negative health effects from chronic or repeated cycles of body weight reduction.

In a rapidly expanding martial arts industry in the US, there have been several reports on sexual assault. Still, no systematic and first-hand documentation on this issue has been completed. In Norway the same increase in popularity of material arts are noticed, an interest also seen among females. With regards to the limited knowledge on exercise practice, eating routines and health symptoms in female material art athletes, this study aims to expand this. By relying on a cross sectional cohort design with systematic registration of outcomes, this study also aim to expand on current limited knowledge on experiences of sexual harassment among females in material arts.

All females aged 16-35 practicing material arts in Oslo (Norway) at the time of recruitment (september-december 2020) will be invited (estimated to be between 200-300 athletes). All participants will receive information on the aim of this study, and must sign informed consent before participation. All data will be measured once per athlete.

ELIGIBILITY:
Inclusion Criteria:

* martial art athlete
* living and training in Oslo-area (main capital) in Norway

Exclusion Criteria:

* not matching sex, age or sport criteria

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Female martial art athletes within sports of boxsing, thaiboxing, kickboxsing, judo, jui jitsu, brasilian jui jitsu, submission wrestling, mixed martial arts, taekwondo og karate.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Low energy availability for females questionnaire (LEAF-Q) | Autumn 2020
  Evaluating intensity in symptoms of low energy availability, with one general score, one subscale measuring symptoms of menstrual irregularities, and one subscale measuring symptoms of gastrointestinal dysfunction; the three scales having cut-off scores of ≥8 , ≥4 and ≥2, with higher scorings indicating higher clinical severity.
Eating disorder examination questionnaire (EDE-q) | Autumn 2020
  Measuring symptoms of eating disorders and frequency of eating disordered behavior, resulting in one total score, and four subscales (figure concern, weight concern, eating concern and eating restriction). A total score of ≥2.5 indicates high probability of having an eating disorder. Additionally, the scales measures frequency of disordered eating behavior, for which ≥1 episode per week of binge-eating and/or ≥1 episode per week of purging behavior, over a total period of ≥3 months, qualifies for an diagnosis of eating disorder.
Body Weight regulation strategies, selfreported | Autumn 2020
  Reports on methods complied with, to achieve body weight reduction (Predefined answers, including an "other" option)
Body appreciation scale (BAS-2) | Autumn 2020
  Evaluates the level of body appreciation and acceptance. Questionnaire contains 10-items with a Likert scale ranging from 1 (Never) to 5 (Always), with a higher average score indicating a higher level of body appreciation.

SECONDARY OUTCOMES:
Exercise frequency, selfreported according to a designed questionnaire | Autumn 2020
  Information on exercise frequency (number of sessions per week)
Exercise duration, selfreported according to a designed questionnaire | Autumn 2020
  Information on duration of sessions (minutes per session)
Exercise motivation, selfreported according to a designed questionnaire | Autumn 2020
  Information on motivation for material arts (reason for choosing the sport, and what level of performance one aims for)
Exercise program variation, selfreported according to a designed questionnaire | Autumn 2020
  Information on the different physical activities performed (reports number of different sport activities undertaken during a typical week)
Physical activity level, objectively measured | Autumn 2020
  Level of physical activity (counts/minute) objectively measured for seven consecutive days using the ActiGraph accelerometer (ActiGraph GT3x and GT3x+, Actigraph, LCC, Pensacola, Florida, USA)
Four day weighed diet registration; energyintake | Autumn 2020
  Four day diet registration by pictures and detailed notes, for analyses of energyintake.
Four day weighed diet registration; nutrient intake | Autumn 2020
  Four day diet registration by pictures and detailed notes, for nutrient analyses. The outcomes will be analysed for total intake of micronutrients specifically found to be in risk of insufficient intake among young norwegian females (calcium, vit-D, folic acid, iodine) and considering their specific needs due to high levels of physically activity (iron and vitamin C) (all given by mg nutrient consumed)
Experiences of sexual harassment | Autumn 2020
  Questions on experiences of sexual harassment, current experience of such, and frequency of such episodes.
Effects from Covid-19 pandemic on exercise- and eating routines, designed questionnaire | Autumn 2020
  Questions on whether covid-19 changed their normal exercise and diet routines (yes/no), if this related to increased or decreased training volume or change in activity preferences. Additionally, whether the pandemic period has changed their energy intake (increased/decreased).

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Sundgot-Borgen, PhD, Study Director — Norwegian School of Sport Sciences
Locations (1):
- Norwegian school of sport sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Data are kept within the scientific group